CLINICAL TRIAL: NCT00618332
Title: Does the Response to a Nasal Decongestant Test Predict the Outcome to Treatment of Seasonal Allergic Rhinitis With Nasonex?
Brief Title: Can a Nasal Decongestant Test Predict Treatment Outcomes in Seasonal Allergic Rhinitis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 15624B
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 2 weeks of treatment
  Interventions: Drug: mometasone furoate nasal spray
- 2 (Placebo Comparator): 2 weeks of treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mometasone furoate nasal spray — 2 puffs in each nostril once a day for 2 weeks
  Other Names: Nasonex
  Arms: 1
Drug: placebo — 2 puffs in each nostril once a day for 2 weeks
  Other Names: placebo comparator for Nasonex
  Arms: 2

SUMMARY:
We hypothesize that those patients with purely seasonal allergic rhinitis will decongest better than those subjects with another cause contributing to their symptoms. These latter patients will not improve as well on an intranasal steroid as those who decongest well, potentially explaining the 60% response rate in prior studies.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 60 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin or RAST test to grass, trees and/or ragweed antigen.
4. Symptomatic at time of entry into study.

Exclusion Criteria

1. Women of childbearing potential not using the contraception method(s) (Birth control pills, depo Provera, double barrier) as well as women who are pregnant or breastfeeding.
2. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (heart, lung, kidney, neurological, oncologic or liver disease).
3. Use of any other investigational agent in the last 30 days.
4. Absence of nasal symptoms.
5. Smoking.
6. URI at the time of screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Sharma S, Vasnani R, De Tineo M, Du G, Pinto JM, Baroody FM, Naclerio RM. Recruitment factors which affect the outcome of a seasonal allergic rhinitis trial. Allergy Asthma Proc. 2011 Jan-Feb;32(1):55-63. doi: 10.2500/aap.2011.32.3414. PMID 21262099

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate: 2 weeks of treatment
  mometasone furoate nasal spray : 2 puffs in each nostril once a day for 2 weeks
- Placebo: 2 weeks of treatment
  placebo : 2 puffs in each nostril once a day for 2 weeks
Period: Overall Study
Arm/Group | Mometasone Furoate | Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (9.36) | 35 (12) | 33.8 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Global Assessment
Description: Global Assessment: 3=significantly improved, 2=moderately improved,
  1=mildly improved, 0=no change, -1=mildly worse, -2=moderately worse, and -3=significantly worse
Time Frame: at week 2
Population: There were one patient in the Mometasone Furoate group and two patients in the Placebo group with missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 1.7 (1.1) [0 to 3] | 1.4 (1.2) [-1 to 3]
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.372, t-test, 2 sided

2. Secondary Outcome: Changes in RQLQ: Overall
Description: The RQLQ is a disease-specific measure of a patient's quality of life. It includes domains that measure nasal and eye symptoms as well as those of activity, sleep, non-nasal/eye symptoms, practical and emotional measures. A scale of 0-6 is used to record the patient responses, with lower scores reflecting a better quality of life. The average score of each domain is calculated as well as an overall domain score reflecting the average of all scores.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.35 (1.09) | -1.25 (1.09)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.775, t-test, 2 sided

3. Secondary Outcome: Changes in RQLQ: Activity
Description: The RQLQ activity range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.73 (1.64) | -1.55 (1.78)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.737, t-test, 2 sided

4. Secondary Outcome: Changes in RQLQ: Sleep
Description: The RQLQ sleep range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.42 (1.18) | -0.85 (1.05)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.117, t-test, 2 sided

5. Secondary Outcome: Changes in RQLQ: Non-Nasal/Eye
Description: The RQLQ non-nasal/eye range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.11 (1.05) | -1.26 (1.22)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.676, t-test, 2 sided

6. Secondary Outcome: Changes in RQLQ: Practical
Description: The RQLQ practical range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.37 (1.26) | -1.48 (1.54)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.795, t-test, 2 sided

7. Secondary Outcome: Changes in RQLQ: Nasal
Description: The RQLQ nasal range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.54 (1.47) | -1.31 (1.53)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.638, t-test, 2 sided

8. Secondary Outcome: Changes in RQLQ: Emotional
Description: The RQLQ emotional range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Population: There were one patient in the Mometasone Furoate group with a missing value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 19 | 20
units on a scale | -1.05 (1.57) | -0.94 (1.24)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.800, t-test, 2 sided

9. Secondary Outcome: Changes in RQLQ: Eye
Description: The RQLQ eye range: 0-6. Higher scores indicate a worse quality of life.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.36 (1.41) | -1.34 (1.32)
Statistical Analysis 1: Comparison: Mometasone Furoate vs Placebo; Test type: Superiority or Other; p = 0.968, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No